CLINICAL TRIAL: NCT06852118
Title: Efficacy of Adductor Magnus Muscle Plane Injection for Sciatic Nerve Block Versus Subgluteal Approach in Combination with Femoral Nerve Block in Knee Surgeries- a Randomized Control Study.
Brief Title: Using the Adductor Magnus Plain Block As an Innovative Approach for Sciatic Nerve Block for Lower Limb Surgeries.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Gaber Saad (Other)
Responsible Party: Sponsor-Investigator, Mohammed Gaber Saad, Lecturer of anesthesia, intensive care and pain medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anesth-.0435/2024 Med Research
Record Dates: First submitted 2025-02-22; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Adductor Magnus Plain Injection for Sciatic Nerve Block
Keywords: sciatic nerve block; Femoral nerve; Adductor magnus muscle; knee surgeries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AMM Group: Adductor Magnus Muscle Plane approach + Femoral Nerve Blocks (Experimental): Conduct the sciatic nerve block via adductor magnus plain injection. the femoral nerve block will be conducted as well
  Interventions: Procedure: AMM Group: Adductor Magnus Muscle Plane approach + Femoral Nerve Blocks
- SG Group: Sciatic nerve block by sub-gluteal approach + Femoral nerve blocks (Active Comparator): Conduct the sciatic nerve block via sub-gluteal approach. the femoral nerve block will be conducted as well
  Interventions: Procedure: SG Group: Sciatic nerve block by sub-gluteal approach + Femoral nerve blocks

INTERVENTIONS:
Procedure: AMM Group: Adductor Magnus Muscle Plane approach + Femoral Nerve Blocks — In the supine position, the femoral nerve block will be conducted using a high-frequency ultrasound probe to identify the femoral nerve just below the fascia iliaca. After proper sterilization, the needle will be advanced in-plane to inject 15 ml bupivacaine 0.5% around the nerve. After performing the femoral nerve block, the adductor magnus muscle plane block will be performed using a low-frequency ultrasound probe positioned 6 cm distal to the inguinal crease to identify the sartorius muscle, femoral artery, femoral vein, and femoral nerve on the deep side of the sartorius muscle, the probe will be slide by about 2-2.5 cm distally, where we could identify the plane between the adductor magnus and the semimembranosus muscles, and after proper sterilization, the needle will be slowly advanced until the needle tip is close to the posterior surface of the AMM, 20 mL of bupivacaine 0.5% will be injected while observing fluid distribution under the posterior surface of the AMM, Then GA.
  Arms: AMM Group: Adductor Magnus Muscle Plane approach + Femoral Nerve Blocks
Procedure: SG Group: Sciatic nerve block by sub-gluteal approach + Femoral nerve blocks — While the patient is in the supine position, the femoral nerve block will be conducted using a high-frequency ultrasound probe to identify a cross-sectional view of the femoral nerve just below the fascia iliaca. After proper sterilization, the needle will be advanced in-plane to inject 15 ml bupivacaine 0.5% around the nerve. the patient will be turned on their sides with the operative side uppermost and flexed, the sub-gluteal sciatic nerve will be identified using a low-frequency probe, and then the same needle will be advanced the in-plane to inject 20 ml bupivacaine 0.5% around the nerve., then GA will be conducted as the other group
  Arms: SG Group: Sciatic nerve block by sub-gluteal approach + Femoral nerve blocks

SUMMARY:
the goal of this clinical trial is to compare the efficacy of adductor magnus muscle plane injection as an approach for sciatic nerve block to sub-gluteal approach in combination with femoral nerve blocks as perioperative analgesia in knee surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anaesthesiologists) Physical Status I-III.
* Patients who consent to receive regional anesthesia.

Exclusion Criteria:

* Patients with a history of allergy to local anesthetics.
* Pre-existing neurological deficits in the lower extremities.
* Coagulopathy or anticoagulation therapy that cannot be safely discontinued.
* Infection at the site of block injection.
* Severe obesity (BMI > 40).
* Patients with contraindications to regional anesthesia.
* peripheral neuropathy.
* Psychiatric disorders and communication difficulties.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of sciatic sensory block | At 30 minutes after the block
  It will be assessed by evaluating the sharp sensation with pinprick testing, and the presence or loss of cold-warm feeling as (2 for normal sensory perception, 1 for loss of cold-warm feeling, and 0 for loss of pinprick sensation) for ciatic in the sole of foot.
Assessment of sciatic motor block | At 30 minutes after the block
  Sciatic block will be evaluated by the motion of the foot and ankle joint (3 for normal movement, 2 for unable to push or flex the foot against external resistance, 1 for unable to push or flex the foot against gravity and 0 for no motion

SECONDARY OUTCOMES:
Postoperative pain scores | At 1, 6, 12, and 24 hours post-operative
  Using the Visual Analog Scale (VAS)
The onset of sciatic sensory blockades | Every 3 minutes with maximum time 30 minutes (if no changes within 30 min the patient will be excluded from the study)
  Time in minutes from removing of the local anesthesia needle to the start of sensory changes
The duration of the sciatic nerve block procedure | during sciatic nerve block conduction
  the time in minutes from the start of the sonographic examination for the sciatic nerve block until local anaesthetic administration.
Visibility scores for the sciatic nerve | during sciatic nerve block using sub gluteal approach conduction
  using a 6-point visibility scale: 0: No nerve was identified
  1. Nerve identified with a high probability
  2. Nerve identified but most of it was not visible
  3. Nerve identified and more than 50% of its borders were precisely distinguished from the surrounding structures
  4. Nerve completely visible but fascicles poorly defined
  5. Nerve completely visible and multiple fascicles identifiable
Visibility scores for Adductor magnus muscle (AMM) | during sciatic nerve block using adductor magnus muscle plain block conduction
  using a 6-point visibility scale for AMM: 0: No muscle was identified
  1. Muscle identified with a high probability
  2. Muscle identified but most of it was not visible
  3. Muscle identified and more than 50% of its epimysium were precisely distinguished from the surrounding structures
  4. Muscle completely visible but perimysium poorly defined
  5. Muscle completely visible and multiple perimysium identifiable
Patient satisfaction | Before the patient discharge
  Using 4 degrees scale: excellent, good, sufficient, insufficient
The onset of the Sciatic motor block | Every 3 minutes with maximum time 30 minutes (if no changes within 30 min the patient will be excluded from the study)
  Time in minutes from removing of the local anesthesia needle to the start of motor changes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculity of medicine - Al-Azhar University hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ben-David B, Schmalenberger K, Chelly JE. Analgesia after total knee arthroplasty: is continuous sciatic blockade needed in addition to continuous femoral blockade? Anesth Analg. 2004 Mar;98(3):747-9, table of contents. doi: 10.1213/01.ane.0000096186.89230.56. PMID 14980931
- [Background] Shanthanna H, Singh B, Guyatt G. A systematic review and meta-analysis of caudal block as compared to noncaudal regional techniques for inguinal surgeries in children. Biomed Res Int. 2014;2014:890626. doi: 10.1155/2014/890626. Epub 2014 Aug 5. PMID 25162033
- [Background] Wang L, Qu Y, Deng Y, Li J, Liu Y, Wu C. Evaluation of a New Method of Sciatic Nerve Block: A Prospective Pilot Study. J Pain Res. 2023 Jun 16;16:2091-2099. doi: 10.2147/JPR.S404489. eCollection 2023. PMID 37346396